CLINICAL TRIAL: NCT03828552
Title: Parents' Experience of Their Children Stay in a Pediatric Intensive Care Unit.
Acronym: VECUREA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0700
Record Dates: First submitted 2019-01-25; First posted 2019-02-04 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Intensive Care Unit Syndrome
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Parents will be recruited in a Pediatric Resuscitation Department of the Mother and Child Hospital for 3 months. The doctor taking care of a child and his parents meeting the eligibility criteria will distribute, during the stay, a questionnaire accompanied by a pre-stamped envelope to the two parents not opposing the study.
  A phone call and / or an email reminder by the intern in the month of the exit will invite each parent to return the questionnaire.
  The completed questionnaire will be mailed back by the parents using the pre-stamped envelope.

SUMMARY:
Children recovered in pediatric intensive care unit (PICU) suffer from severe conditions, sometimes life-threatening. Thus, priority is given to urgent somatic care, children medicalization is strong, invasive technics have to be used, and medical monitoring is close.

A stay in PICU often leaves a painful memory to the child and family, and can lead to psychological morbidity such as post-traumatic stress disease.

This study aims to assess parents' experience during their child hospitalization in PICU, and the impact of this stay on the entire family in the following month.

ELIGIBILITY:
Inclusion Criteria:

* Parent (mother or /and father) of a recovered child in PICU.
* No limit of age, disease or admission mode.
* First stay in PICU, for at least a 3 days stay.
* Parents having been informed and having accepted the participation in the study.

Exclusion Criteria:

* Death of the child during the stay in PICU or during the month following the discharge from PICU
* Non-fluent french speakers/readers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parent (mother or /and father) of a recovered child in the PICU for at least 3 days, for a first stay, without limit of age, disease or admission mode.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Analyse qualitatively the parents'experience during the PICU stay of their child | 1 month
  Analysis of french written answers on a feedback form of about 10 pages (free written answers or Likert scale)
Assessment of the impact on the family of this PICU stay of their child | 1 month
  Analysis of french written answers on a feedback form of about 10 pages (free written answers or Likert scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric intensive care unit of Women-Mother-Children Hospital, Bron, France

IPD SHARING:
Plan to Share IPD: No